CLINICAL TRIAL: NCT01255163
Title: A Pilot Study of Exendin-4 in Alzheimer s Disease
Brief Title: A Pilot Clinical Trial of Exendin-4 in Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: AstraZeneca withdrew support for the study.
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100423; 10-AG-0423
Record Dates: First submitted 2010-12-04; First posted 2010-12-07 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Alzheimer's; Brain insulin resistance; Diabetes
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo-controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study with code kept by NIA Pharmacist who did not share with Investigators and had no interaction with participants and caregivers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exendin-4 (Experimental): Exenatide 5 mcg or 10 mcg SC twice daily
  Interventions: Drug: Exendin-4 SC
- Placebo (Placebo Comparator): Placebo SC twice daily
  Interventions: Drug: Placebo SC

INTERVENTIONS:
Drug: Exendin-4 SC — Exenatide 5 mcg or 10 mcg SC twice daily
  Other Names: Exenatide SC
  Arms: Exendin-4
Drug: Placebo SC — Placebo SC twice daily
  Other Names: Placebo SC twice daily
  Arms: Placebo

SUMMARY:
Background:

Exendin-4 (or Exenatide) is a medication currently used to treat diabetes that has shown promising results in animal and cellular models of Alzheimer's disease. It is possible that Exendin-4 may be a treatment for Alzheimer's disease, which involves the gradual deterioration and death of neurons. Researchers are interested in studying the safety and comparing the effects of Exendin-4 with placebo on cognitive performance, clinical progression of dementia, various chemicals measured in blood and cerebrospinal fluid, and brain MRI, in individuals with early-stage Alzheimer's disease or mild cognitive impairment.

Objectives:

To determine the safety and tolerability of twice daily administration of Exendin-4, as well as to acquire preliminary evidence for effects on cognitive performance, clinical progression of dementia, various chemicals measured in blood and cerebrospinal fluid, and brain MRI, in individuals with early-stage Alzheimer's disease or mild cognitive impairment.

Eligibility:

Individuals at least 60 years of age who have objective evidence of early-stage Alzheimer's disease or mild cognitive impairment in screening testing.

Design:

* Participants will be screened.
* Following the telephone screening, two in-person screening visits to determine eligibility.
* The screening visit will involve a medical history and neurological examination, tests of memory and cognition, a lumbar puncture, collection of blood and saliva samples, and brain Magnetic Resonance Imagine (MRI) studies. Participants will be required to appoint a Durable Power of Attorney for research and medical care during this protocol.
* Eligible participants will be divided into two groups (double-blind randomization). One group will receive Exendin-4 SC twice daily, and the other will receive a placebo. Participants will keep a medication diary and will be scheduled for additional study visits 1 and 2 weeks after the start of the treatment.
* Participants will have regular followup visits with blood tests, cognitive tests, imaging studies, and other examinations 6, 12, and 18 months after the start of the treatment. Another lumbar puncture may be performed optionally at the 18-month followup visit.

DETAILED DESCRIPTION:
Objective: Exendin-4 (or exenatide) is a medication currently used in the treatment of diabetes mellitus (DM). Exendin-4 has generated promising results as an agent protecting neurons from a number of assaults both in the laboratory and in studies on animals. Specifically, there is pre-clinical evidence that Exendin-4 may be a treatment for Alzheimer's disease (AD). Based on these facts, we conducted a pilot Phase II double blind randomized placebo-controlled clinical study to assess the safety and provide proof of concept for exendin-4 treatment in early Alzheimer's disease (AD), by demonstrating a response of disease biomarkers to the intervention. Our main hypothesis is that long-term administration of Exendin-4 in participants with amnestic MCI/early AD in FDA-approved doses is safe and will induce a change over time in AD biomarkers. Subject population: We intend to screen up to 100 potential participants in order to ensure that at least 40 participants (enrolled based on a clinical diagnosis of amnestic MCI/early AD and Cerebrospinal Fluid (CSF) biomarker evidence of AD) will be enrolled into treatment and complete the study. Design: Enrolled participants will be randomly assigned into one of two groups (Exendin-4 vs. Placebo) and will be followed at regular intervals for 18 months. Outcome measures: Safety and tolerability will be the primary outcomes. In addition, we will measure and assess the change over time of a number of exploratory outcomes with the intervention, including CSF and plasma biomarkers (such as CSF A42, tau, p181-tau and plasma A42/A40), cognitive performance measures (such as the Alzheimer's Disease Assessment scale, cognitive sub-scale, and other tests), clinical progression of dementia measures (such as the Clinical Dementia Rating scale sum-of-boxes), volumetric changes on structural brain MRI and changes in resting fMRI. All research will be performed on the National Institute on Aging (NIA) Clinical Research Unit located on the 5th floor of Harbor Hospital.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age > 60
* Clinical Dementia Rating (global CDR) of 0.5 or 1. Memory box score must be at least 0.5.
* Mini Mental Status Exam (MMSE) > 20
* Clinical diagnosis of (amnestic or mixed) MCI or early AD and Memory deficit on neuropsychological or clinical testing.
* Hamilton Depression Scale score of less than or equal to 12 on the 17-item scale
* CSF A beta 42 < 192 (+- 10%) pg/ml (given an intra-subject laboratory variability ~ 10%)
* Medications stable for at least 4 weeks prior to screening. In particular:

  * Participants may take stable doses of antidepressants, chronic anxiolytics or sedative hypnotics, if started at least 4 weeks or longer prior to screening
  * Cholinesterase inhibitors and/or memantine are allowable, if started at least 4 weeks prior to screening
  * Participants will not be asked to discontinue medications without permission from their primary care provider (PCP) or specialist.
* Fluency in English
* At the time of enrollment, participants must have the ability to provide informed consent and make health care decisions.
* An informant or caregiver who has frequent contact with the participant (e.g. an average of 10 hours per week or more) must be appointed to serve as Durable Power of Attorney (DPA) for research and medical care at NIA, accompany the participant to clinic visits and provide historical information regarding the participant s cognitive status, and assist participants with/administer injections of the investigational medication.
* Good general health with no additional disease states that could interfere with the study.

EXCLUSION CRITERIA:

* Other significant neurological disease of the Central Nervous System (such as Parkinson s disease, atypical Parkinsons disease, Multi-infarct Dementia, Frontotemporal Dementia, Huntington s disease, Normal Pressure Hydrocephalus, brain tumor, Progressive Supranuclear Palsy, Epilepsy, Subdural Hematoma or Multiple Sclerosis)
* A history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities
* Positive RPR or HIV
* Abnormal PT/PTT and INR (1.5 standard deviation over the upper normal limit) increasing the risk for LP related bleeding/hematoma; platelet count <100,000/microliters.
* Anti-coagulant therapy (such as coumadin). Aspirin up to 325 is allowed.
* Investigators unable to obtain CSF, failure of Lumbar Puncture after a limited number of unsuccessful attempts).
* History of psychiatric disease with significant impairment in thought processes (e.g. schizophrenia, bipolar disease, psychosis). Participants who develop psychiatric conditions necessitating treatment after their enrollment will not be dropped from the study. The high incidence of late-onset depression and anxiety among individuals with MCI and AD requires that participants with depression, and/or anxiety should not be excluded from the cohort to maintain the ecological validity of the results.
* Current abuse of alcoholic beverages (> 7 in women and >14 in men) or substance abuse.
* Known diagnosis of diabetes at the time of enrollment or new diagnosis of diabetes based on the findings of elevated fasting blood glucose (= or >126 mg/dl) and/or the oral glucose tolerance test at screening (>200 mg/dl at two hours).
* Severe renal impairment (creatinine clearance <30 ml/min) or end-stage renal disease. Individuals with moderate renal impairment (creatinine clearance 30 to 50 ml/min) may be enrolled in the study, but their BUN and Creatinine will be monitored during each visit after drug initiation and extra safety visits will be conducted at 3, 9, and 15 months.
* Current or previous treatment with Exendin-4 (Exenatide, trade name Byetta.)
* History of pancreatitis, active upper GI, hepatic or gallbladder disease
* Personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia syndrome type 2
* History of repeated hypoglycemia
* Body mass index (BMI) < 18 on enrollment (given the expected weight loss caused by Exendin-4 and dementia). In the BLSA, participants with age > 65 had a mean BMI of 25.8 with SD of 3.9 Exendin-4 has been shown to cause an average 5.3 kg weight loss, with 95% CI: 6 to 4.5 kg (126).
* Allergy to Exendin-4 or to substances in the injection pen (metacresol, mannitol, glacial acetic acid, sodium acetate trihydrate, water for injection).
* Participation in other studies of investigational treatments for Alzheimer s disease in the last year.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-11-21; Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios I Kapogiannis, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute on Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kapogiannis D, Mattson MP. Disrupted energy metabolism and neuronal circuit dysfunction in cognitive impairment and Alzheimer's disease. Lancet Neurol. 2011 Feb;10(2):187-98. doi: 10.1016/S1474-4422(10)70277-5. Epub 2010 Dec 10. PMID 21147038
- [Background] Bomfim TR, Forny-Germano L, Sathler LB, Brito-Moreira J, Houzel JC, Decker H, Silverman MA, Kazi H, Melo HM, McClean PL, Holscher C, Arnold SE, Talbot K, Klein WL, Munoz DP, Ferreira ST, De Felice FG. An anti-diabetes agent protects the mouse brain from defective insulin signaling caused by Alzheimer's disease- associated Abeta oligomers. J Clin Invest. 2012 Apr;122(4):1339-53. doi: 10.1172/JCI57256. PMID 22476196
- [Derived] Liu QR, Zhu M, Chen Q, Mustapic M, Kapogiannis D, Egan JM. Novel Hominid-Specific IAPP Isoforms: Potential Biomarkers of Early Alzheimer's Disease and Inhibitors of Amyloid Formation. Biomolecules. 2023 Jan 13;13(1):167. doi: 10.3390/biom13010167. PMID 36671553
- [Derived] Mullins RJ, Mustapic M, Chia CW, Carlson O, Gulyani S, Tran J, Li Y, Mattson MP, Resnick S, Egan JM, Greig NH, Kapogiannis D. A Pilot Study of Exenatide Actions in Alzheimer's Disease. Curr Alzheimer Res. 2019;16(8):741-752. doi: 10.2174/1567205016666190913155950. PMID 31518224
- [Derived] Muscogiuri G, DeFronzo RA, Gastaldelli A, Holst JJ. Glucagon-like Peptide-1 and the Central/Peripheral Nervous System: Crosstalk in Diabetes. Trends Endocrinol Metab. 2017 Feb;28(2):88-103. doi: 10.1016/j.tem.2016.10.001. Epub 2016 Oct 27. PMID 27871675
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-AG-0423.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between 10/5/2010 and 7/25/2016. A total of 57 participants signed informed consent to undergo screening procedures. Of those, 28 qualified, 1 withdrew prior to randomization, 27 were randomized to exenatide or placebo, and 18 completed the study.
Pre-assignment Details: The study includes a baseline visit to determine eligibility. Therefore, 57 participants were enrolled (i.e. signed informed consent prior to screening). Of those, 28 qualified, 1 withdrew prior to randomization, 27 were randomized to exenatide or placebo, and 18 completed the study.
Period: Overall Study
Arm/Group | Exendin-4 | Placebo
Started | 13 | 14
Completed | 9 | 9
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 0 | 2
Not completed — AstraZeneca stopped support of the study | 1 | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes 27 participants who underwent randomization and received at least one dose of experimental medication. Of those 27, we have at least one outcome measure (i.e. at least the 6 months follow-up data point) for 21 participants. Of those 21, 18 completed the study (i.e. reached 18 months).
Groups:
- Total: Total of all reporting groups
Arm/Group | Exendin-4 | Placebo | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.46 (7.137) | 74.64 (7.034) | 72.63 (7.265)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27
Cerebrospinal fluid amyloid-beta 42 (CSF Abeta42) [Mean (Standard Deviation); unit: pg/dl] — Measured in CSF using Luminex xMAP technology and INNO-BIA Alz Bio3 kits (Research Use Only) provided by Fujirebio
  pg/dl | 158.85 (43.619) | 158.86 (33.558) | 158.85 (37.963)
Mini Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Scale range: 0 - 30 points (higher is better)
  units on a scale | 25.85 (3.997) | 24.64 (5.198) | 25.22 (4.61)
Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog70) [Mean (Standard Deviation); unit: units on a scale] — Alzheimer's dementia scale cognitive sub-scale range: 0 - 70 points (higher is worse)
  units on a scale | 14.46 (6.654) | 13.64 (6.879) | 14.04 (6.653)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index defined as a person's weight in kilograms (kg) divided by his or her height in meters squared.
  kg/m^2 | 26.631 (3.3673) | 26.85 (5.2611) | 26.744 (4.3687)
Fasting glucose [Mean (Standard Deviation); unit: mg/dl] | 94.92 (8.311) | 90.14 (9.206) | 92.44 (8.954)
Fasting insulin [Mean (Standard Deviation); unit: uIU/ml] | 8.53 (4.4337) | 8.1 (4.5361) | 8.254 (4.4628)
Cerebrospinal fluid phospho181-tau (CSF p181-tau) [Mean (Standard Deviation); unit: pg/dl] — Measured in CSF using Luminex xMAP technology and INNO-BIA Alz Bio3 kits (Research Use Only) provided by Fujirebio
  pg/dl | 56.62 (34.606) | 40.64 (16.137) | 48.33 (27.369)
Cerebrospinal fluid (CSF) Total Tau [Mean (Standard Deviation); unit: pg/dl] — Measured in CSF using Luminex xMAP technology and INNO-BIA Alz Bio3 kits (Research Use Only) provided by Fujirebio
  pg/dl | 90.38 (53.053) | 70.64 (22.802) | 80.15 (40.744)
Clinical Dementia Rating (CDR) global score [Mean (Standard Deviation); unit: units on a scale] — Clinical Dementia Rating global score range: 0 (no dementia); 0.5 (Mild Cognitive Impairment); 1 (mild dementia); 2 (moderate dementia); 3 (severe dementia). Higher is worse.
  units on a scale | 0.577 (0.2774) | 0.607 (0.2129) | 0.593 (0.2417)
Clinical Dementia Rating (CDR) sum of boxes [Mean (Standard Deviation); unit: units on a scale] — Sum of the Clinical Dementia Rating "boxes" (memory, orientation, judgment and problem solving, community affairs, home and hobbies, personal care). Each box is rated as 0, 0.5, 1, 2 or 3. Range for the sum of boxes is 0 - 18. Higher scores reflect a greater severity of dementia.
  units on a scale | 2.769 (1.775) | 3 (1.7759) | 2.889 (1.745)
Nausea [Count of Participants; unit: Participants] — Nausea reported by participant
  Participants | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Nausea
Description: Tolerability of exenatide (nausea is the most common expected adverse event of exenatide)
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Exendin-4 | Placebo
Number analyzed (Participants) | 13 | 14
Participants | 5 | 0
Statistical Analysis 1: Comparison: Exendin-4 vs Placebo; Test type: Other; p = 0.016, Fisher Exact — threshold for significance (p < 0.05)

2. Secondary Outcome: Mini Mental State Examination (MMSE)
Description: Scale range: 0 - 30 points (higher is better)
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exendin-4 | Placebo
Number analyzed (Participants) | 13 | 14
units on a scale | 23.11 (6.009) | 23.11 (5.011)
Statistical Analysis 1: Comparison: Exendin-4 vs Placebo; Test type: Other; p = 0.098, Mixed Models Analysis — Threshold for statistical significance p < 0.05. Type III Tests of Fixed Effects Group * VisitLong F (6, 52.008) = 1.902, p = 0.098; Repeated measures mixed model with Repeated Factor (Visit Long: baseline, 6, 12, 18 months), Fixed Factors (Group,VisitLong, Sex) and Covariate (Age); MIXED MMSE.tot BY Group Sex VisitLong WITH Age * CRITERIA=CIN(95) MXITER(100) MXSTEP(10) SCORING(1) SINGULAR(0.000000000001) HCONVERGE(0, ABSOLUTE) LCONVERGE(0, ABSOLUTE) PCONVERGE(0.000001, ABSOLUTE) * FIXED=Group Sex Age Group*VisitLong | SSTYPE(3) * METHOD=REML * PRINT=SOLUTION * REPEATED=VisitLong | SUBJECT(SubjectID) COVTYPE(AR1) * EMMEANS=TABLES(Group) COMPARE ADJ(BONFERRONI) * EMMEANS=TABLES(Sex) COMPARE ADJ(BONFERRONI) * EMMEANS=TABLES(Group*VisitLong) COMPARE(Group) ADJ(BONFERRONI) * EMMEANS=TABLES(Group*VisitLong) COMPARE(VisitLong) ADJ(BONFERRONI)

3. Secondary Outcome: Alzheimer's Disease Assessment Scale-cognitive Subscale (ADAS-cog70)
Description: Alzheimer's dementia scale cognitive sub-scale range: 0 - 70 points (higher is worse)
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exendin-4 | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | 16 (8.588) | 17.78 (8.643)
Statistical Analysis 1: Comparison: Exendin-4 vs Placebo; Test type: Other; p = 0.295, Mixed Models Analysis — Threshold for statistical significance p < 0.05. Type III Tests of Fixed Effects for Group*VisitLong F (6, 52.281) = 1.254, p = 0.295; [statistical method as in outcome 2, analysis 1]; MIXED ADAS70 BY Group Sex VisitLong WITH Age * CRITERIA=CIN(95) MXITER(100) MXSTEP(10) SCORING(1) SINGULAR(0.000000000001) HCONVERGE(0, ABSOLUTE) LCONVERGE(0, ABSOLUTE) PCONVERGE(0.000001, ABSOLUTE) * FIXED=Group Sex Age Group*VisitLong | SSTYPE(3) * METHOD=REML * PRINT=SOLUTION * REPEATED=VisitLong | SUBJECT(SubjectID) COVTYPE(AR1) * EMMEANS=TABLES(Group) COMPARE ADJ(BONFERRONI) * EMMEANS=TABLES(Sex) COMPARE ADJ(BONFERRONI) * EMMEANS=TABLES(Group*VisitLong) COMPARE(Group) ADJ(BONFERRONI) * EMMEANS=TABLES(Group*VisitLong) COMPARE(VisitLong) ADJ(BONFERRONI)

4. Secondary Outcome: Clinical Dementia Rating (CDR) Global Score
Description: Clinical Dementia Rating global score range: 0 (no dementia); 0.5 (Mild Cognitive Impairment); 1 (mild dementia); 2 (moderate dementia); 3 (severe dementia). Higher is worse.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exendin-4 | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | 0.889 (0.6509) | 0.833 (0.5)
Statistical Analysis 1: Comparison: Exendin-4 vs Placebo; Test type: Other; p = 0.141, Mixed Models Analysis — Threshold for statistical significance p < 0.05. Type III Tests of Fixed Effects Group * VisitLong F (6, 47.485) = 1.704, p = 0.141; [statistical method as in outcome 2, analysis 1]; MIXED CDR BY Group Sex VisitLong WITH Age CRITERIA=CIN(95) MXITER(100) MXSTEP(10) SCORING(1) SINGULAR(0.000000000001) HCONVERGE(0, ABSOLUTE) LCONVERGE(0, ABSOLUTE) PCONVERGE(0.000001, ABSOLUTE) FIXED=Group Sex Age Group*VisitLong | SSTYPE(3) METHOD=REML PRINT=SOLUTION REPEATED=VisitLong | SUBJECT(SubjectID) COVTYPE(AR1) EMMEANS=TABLES(Group) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Sex) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(Group) ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(VisitLong) ADJ(BONFERRONI)

5. Secondary Outcome: Clinical Dementia Rating (CDR) Sum of Boxes
Description: Sum of the Clinical Dementia Rating "boxes" (memory, orientation, judgment and problem solving, community affairs, home and hobbies, personal care). Each box is rated as 0, 0.5, 1, 2 or 3. Range for the sum of boxes is 0 - 18. Higher scores reflect a greater severity of dementia.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exendin-4 | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | 4.778 (4.0782) | 4.5 (2.3318)
Statistical Analysis 1: Comparison: Exendin-4 vs Placebo; Test type: Other; p = 0.031, Mixed Models Analysis — Threshold for statistical significance p < 0.05. Type III Tests of Fixed Effects: Group * VisitLong F (6, 51.955) = 2.553, p = 0.031. Univarate Exendin-4 F(3, 51.386) = 2.734, p = 0.053. Pairwise for Exendin-4, baseline vs. 18 months (p = 0.035); [statistical method as in outcome 2, analysis 1]; MIXED CDR.sob BY Group Sex VisitLong WITH Age CRITERIA=CIN(95) MXITER(100) MXSTEP(10) SCORING(1) SINGULAR(0.000000000001) HCONVERGE(0, ABSOLUTE) LCONVERGE(0, ABSOLUTE) PCONVERGE(0.000001, ABSOLUTE) FIXED=Group Sex Age Group*VisitLong | SSTYPE(3) METHOD=REML PRINT=SOLUTION REPEATED=VisitLong | SUBJECT(SubjectID) COVTYPE(AR1) EMMEANS=TABLES(Group) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Sex) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(Group) ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(VisitLong) ADJ(BONFERRONI)

6. Secondary Outcome: Cerebrospinal Fluid (CSF) Total Tau
Description: Total Tau measured in CSF using Luminex xMAP technology and INNO-BIA Alz Bio3 kits (Research Use Only) provided by Fujirebio
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: pg/dl
Arm/Group | Exendin-4 | Placebo
Number analyzed (Participants) | 9 | 9
pg/dl | 86.57 (37.434) | 70.75 (33.148)
Statistical Analysis 1: Comparison: Exendin-4 vs Placebo; Test type: Other; p = 0.703, Mixed Models Analysis — Threshold for statistical significance p < 0.05. Type III Tests of Fixed Effects Group * VisitLong F (2, 15.251) = 0.360, p = 0.703; Repeated measures mixed model with Repeated Factor (Visit Long: baseline,18 months), Fixed Factors (Group,VisitLong, Sex) and Covariate (Age); MIXED TAU BY Group Sex VisitLong WITH Age CRITERIA=CIN(95) MXITER(100) MXSTEP(10) SCORING(1) SINGULAR(0.000000000001) HCONVERGE(0, ABSOLUTE) LCONVERGE(0, ABSOLUTE) PCONVERGE(0.000001, ABSOLUTE) FIXED=Group Sex Age Group*VisitLong | SSTYPE(3) METHOD=REML PRINT=SOLUTION REPEATED=VisitLong | SUBJECT(SubjectID) COVTYPE(AR1) EMMEANS=TABLES(Group) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Sex) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(Group) ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(VisitLong) ADJ(BONFERRONI)

7. Secondary Outcome: Cerebrospinal Fluid phospho181-tau (CSF p181-tau)
Description: p-181-Tau measured in CSF using Luminex xMAP technology and INNO-BIA Alz Bio3 kits (Research Use Only) provided by Fujirebio
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: pg/dl
Arm/Group | Exendin-4 | Placebo
Number analyzed (Participants) | 9 | 9
pg/dl | 54.57 (32.893) | 44.25 (19.739)
Statistical Analysis 1: Comparison: Exendin-4 vs Placebo; Test type: Other; p = 0.845, Mixed Models Analysis — Threshold for statistical significance p < 0.05. Type III Tests of Fixed Effects Group * VisitLong F (2, 15.828) = 0.170, p = 0.845; [statistical method as in outcome 6, analysis 1]; MIXED pTAU BY Group Sex VisitLong WITH Age CRITERIA=CIN(95) MXITER(100) MXSTEP(10) SCORING(1) SINGULAR(0.000000000001) HCONVERGE(0, ABSOLUTE) LCONVERGE(0, ABSOLUTE) PCONVERGE(0.000001, ABSOLUTE) FIXED=Group Sex Age Group*VisitLong | SSTYPE(3) METHOD=REML PRINT=SOLUTION REPEATED=VisitLong | SUBJECT(SubjectID) COVTYPE(AR1) EMMEANS=TABLES(Group) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Sex) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(Group) ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(VisitLong) ADJ(BONFERRONI)

8. Secondary Outcome: Cerebrospinal Fluid Amyloid-beta 42 (CSF Abeta42)
Description: Abeta42 peptide measured in CSF using Luminex xMAP technology and INNO-BIA Alz Bio3 kits (Research Use Only) provided by Fujirebio
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: pg/dl
Arm/Group | Exendin-4 | Placebo
Number analyzed (Participants) | 9 | 9
pg/dl | 177.43 (70.720) | 176.38 (30.528)
Statistical Analysis 1: Comparison: Exendin-4 vs Placebo; Test type: Other; p = 0.018, Mixed Models Analysis — Type III Tests of Fixed Effects: Group * VisitLong F (2, 16.614) = 5.142, p = 0.018. Univariate tests: Placebo F(1, 16.595) = 4.138, p = 0.058; Exendin-4 F(1, 16.595) = 6.262, p = 0.022. Pairwise for Exendin-4, baseline vs. 18 months (p = 0.022); [statistical method as in outcome 6, analysis 1]; MIXED Ab42 BY Group Sex VisitLong WITH Age CRITERIA=CIN(95) MXITER(100) MXSTEP(10) SCORING(1) SINGULAR(0.000000000001) HCONVERGE(0, ABSOLUTE) LCONVERGE(0, ABSOLUTE) PCONVERGE(0.000001, ABSOLUTE) FIXED=Group Sex Age Group*VisitLong | SSTYPE(3) METHOD=REML PRINT=SOLUTION REPEATED=VisitLong | SUBJECT(SubjectID) COVTYPE(AR1) EMMEANS=TABLES(Group) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Sex) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(Group) ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(VisitLong) ADJ(BONFERRONI)

9. Secondary Outcome: Body Mass Index (BMI)
Description: Body Mass Index defined as a person's weight in kilograms (kg) divided by his or her height in meters squared.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Exendin-4 | Placebo
Number analyzed (Participants) | 9 | 9
kg/m^2 | 25.867 (3.6284) | 25.789 (4.6023)
Statistical Analysis 1: Comparison: Exendin-4 vs Placebo; Test type: Other; p = 0.009, Mixed Models Analysis — Type III Tests of Fixed Effects: Group * VisitLong F (8, 72.603) = 2.816, p = 0.009. Univarate Exendin-4 F(4, 72.944) = 4.834, p = 0.002. Pairwise comparisons for Exendin-4 showed a decrease in BMI baseline vs. 6 months (p = 0.029); [statistical method as in outcome 2, analysis 1]; MIXED BMI BY Group Sex VisitLong WITH Age CRITERIA=CIN(95) MXITER(100) MXSTEP(10) SCORING(1) SINGULAR(0.000000000001) HCONVERGE(0, ABSOLUTE) LCONVERGE(0, ABSOLUTE) PCONVERGE(0.000001, ABSOLUTE) FIXED=Group Sex Age Group*VisitLong | SSTYPE(3) METHOD=REML PRINT=SOLUTION REPEATED=VisitLong | SUBJECT(SubjectID) COVTYPE(AR1) EMMEANS=TABLES(Group) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Sex) COMPARE ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(Group) ADJ(BONFERRONI) EMMEANS=TABLES(Group*VisitLong) COMPARE(VisitLong) ADJ(BONFERRONI)

ADVERSE EVENTS:
Time Frame: Up to 18 months
Description: Description of AEs according to clinicaltrials.gov definitions
Arm/Group | Exendin-4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/14
Other Adverse Events (participants affected / at risk) | 13/13 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exendin-4 (N=13) | Placebo (N=14)
Myocardiac Infarction (Cardiac disorders) | 1 (1) | 0 (0) — Myocardiac Infarction treated with cardiac stent placement
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Lung cancer diagnosed after pathological fracture 2 days after starting experimental drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exendin-4 (N=13) | Placebo (N=14)
Nausea (Gastrointestinal disorders) | 5 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 — GERD
Lower abdominal pain (Gastrointestinal disorders) | 1 | 0 — Mild lower abdominal pain (all causes)
Pancreatic enzyme elevation (Gastrointestinal disorders) | 2 | 2 — Asymptomatic elevation (over the upper normal limit) in serum amylase (and/or pancreatic-specific amylase) and/or serum lipase
Diarrhea (Gastrointestinal disorders) | 3 | 1 — Mild intermittent diarrhea (all causes)
Loss of appetite/weight loss (Metabolism and nutrition disorders) | 4 | 0 — Loss of appetite leading to weight loss > 5 lb
Hypoglycemia symptoms (Metabolism and nutrition disorders) | 3 | 2 — Mild episodic symptoms consistent with hypoglycemia and relieved by meal (episodic fatigue and/or dizziness and/or lightheadedness and/or diaphoresis and/or nervousness and/or tremulousness). No episodes of severe symptomatic hypoglycemia.
Injection site ecchymosis and pain (Skin and subcutaneous tissue disorders) | 1 | 1
Abnormal kidney function tests (Renal and urinary disorders) | 2 | 2 — Elevation in serum BUN and/or creatinine and/or GFR (over the upper normal limit)
Fatigue (General disorders) | 2 | 0
Thyroid abnormalities (Endocrine disorders) | 1 | 2 — Two participants had changes in thyroid function tests (TSH and/or T4 or FT4) requiring a change in thyroxine regimen. One of them (placebo-treated) had symptomatic hypothyroidism. One placebo participant had thyroid nodules biopsied (benign).
Post lumbar puncture headache (Injury, poisoning and procedural complications) | 3 | 3 — Post lumbar puncture headache (all types). LP takes place during screening and at the 18 month outcome visit. One participant required blood patch after common analgesics and hydration did not provide relief.
Orthopedic injuries (Musculoskeletal and connective tissue disorders) | 2 | 2 — Fractures (all types), lower back pain, strain, etc.
Vomiting (Injury, poisoning and procedural complications) | 1 | 0 — Vomiting from lying flat on the MRI table
Vasovagal syncope (Nervous system disorders) | 2 | 0 — One participant had syncope during the LP procedure (the participant had hiatal hernia and the pressure from bending over caused nausea and vasovagal syncope). Another participant had syncope during a boar ride and experiencing sea sickness.
Lacunar stroke (Nervous system disorders) | 0 | 1 — Asymptomatic subacute lacunar stroke discovered during ER work-up.
Gout (Musculoskeletal and connective tissue disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Allergic conjuctivitis (Eye disorders) | 1 | 0
Floaters (Eye disorders) | 0 | 1
Dyspnea on exertion (Cardiac disorders) | 0 | 1 — Worsening DOE in participant with pre-existing cardiomyopathy

LIMITATIONS AND CAVEATS:
The study was terminated after AstraZeneca withdrew support. Early termination lead to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes